CLINICAL TRIAL: NCT06658821
Title: The Effect of LDL557 on Improving Degenerative Arthritis in the Elderly
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Collaborators: SYNBIO TECH INC. Kaohsiung Taiwan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CS2-24147
Record Dates: First submitted 2024-10-17; First posted 2024-10-26 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Arthritis; Joint Pain
MeSH Terms: conditions — Arthritis; Arthralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LDL557-HK capsule (Experimental): Subjects will take one capsule of the experimental group(LDL557-HK capsule) within 30 minutes before lunch during the experimental period.
  Interventions: Dietary Supplement: LDL557-HK capsule
- Placebo capsule (Placebo Comparator): Subjects will take one placebo capsule within 30 minutes before lunch during the experimental period.
  Interventions: Dietary Supplement: Placebo Capsule

INTERVENTIONS:
Dietary Supplement: LDL557-HK capsule — Subjects will take once a day during the experimental period. one LDL557-HK capsule(Heat-killed Lactobacillus delbrueckii subsp. lactis LDL557 1x10^10cell) within 30 minutes before lunch.
  Arms: LDL557-HK capsule
Dietary Supplement: Placebo Capsule — Subjects will take once a day during the experimental period. one placebo capsule within 30 minutes before lunch.
  Arms: Placebo capsule

SUMMARY:
This project is to conduct a clinical trial of SYNBIO TECH INC.'s LDL557 capsule for joint protection. To understand the improvement of joint discomfort and inflammation after supplementation, we hope to provide an updated choice for modern people's joint protection.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-40 kg/m2;
* Those with early stage degenerative arthritis symptoms judged by X-ray to be Kellgren-Lawrence Grading Scale level 1 or 2, and the physician determines that long-term treatment is not needed or WOMAC score>2.0 or WOMAC total scale score>12 or VAS score ≦6.

Exclusion Criteria:

* Smoking
* alcoholism
* diabetes
* breastfeeding women and pregnant women.
* Those consuming dietary supplements were excluded.
* Those who use non-steroidal anti-inflammatory analgesics and those who have had joint surgery.
* Rheumatoid arthritis.
* Those who have had joint injections within 6 months.
* Those with cardiovascular and cerebrovascular, rheumatoid or mental diseases.
* Patients undergoing cancer treatment.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
WOMAC | Baseline, Week 4, Week 8, and Week 12
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis.
  Higher scores indicate worse pain, stiffness, and functional limitations. The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68).

SECONDARY OUTCOMES:
KOOS | Baseline, Week 4, Week 8, and Week 12
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a questionnaire for patients with knee injuries or osteoarthritis. It helps measure their pain, symptoms, daily activities, sports ability, and quality of life. The scores are converted to 0-100 for each category. A higher score means worse knee problems.
Lequesne's index | Baseline, Week 4, Week 8, and Week 12
  The Lequesne's Index is a questionnaire designed to evaluate the severity of osteoarthritis in the hip or knee. It assesses pain or discomfort during activities, the ability to walk certain distances, and difficulties in daily activities. The total score ranges from 0 to 24, with higher scores indicating more severe symptoms and greater impact on mobility and quality of life.
VAS | Baseline, Week 4, Week 8, and Week 12
  Using the Visual Analogue Scale (VAS) to measure knee pain. Patients rate their pain on a straight line, where 0 means no pain and 10 means the worst pain imaginable. The patient marks a point on the line that represents their pain level, and the score is measured in centimeters or millimeters.
Quality of life (QOL) SF-36 | Baseline, Week 4, Week 8, and Week 12
  The SF-36 questionnaire is widely used to measure perceived health-related quality of life (HRQOL) and daily functioning. It consists of 36 items, which are summarized into two main domains: the Physical Component Summary (PCS) and the Mental Component Summary (MCS).
Kellgren-Lawrence Grade | Baseline and Week 12
  The Kellgren-Lawrence (KL) grading system is a widely used method for classifying the severity of osteoarthritis (OA) based on radiographic findings. It consists of five grades, ranging from 0 to 4 (Normal, Doubtful, Mild, Moderate, Severe)
Joint range of motion assessment | Baseline and Week 12
  Joint range of motion (ROM) assessment evaluates the movement capacity of a joint, focusing on its flexibility and mobility. For the extensor and flexor muscle groups, the assessment measures the degree of joint extension (straightening) and flexion (bending).
Timed Up and Go Test | Baseline and Week 12
  The time taken to rise from a chair, walk 3 meters, turn, return, and sit down will be recorded. Unit of Measure: Seconds (s)
Stair Climb Test | Baseline and Week 12
  Participants will be asked to ascend and descend a standardized flight of stairs, and the time required will be recorded. Unit of Measure: Seconds (s)
Aerobic Capacity | Baseline and Week 12
  Aerobic capacity will be assessed using 6-minute walk test to evaluate endurance. Unit of Measure: Meters (m)
Inflammation assessment | Baseline and Week 12
  Using the ELISA method, measure the serum levels of inflammatory markers, including C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), prostaglandin E2 (PGE2), tumor necrosis factor-alpha (TNF-α), interleukin-1 beta (IL-1β), interleukin-10 (IL-10), matrix metalloproteinase-3 (MMP-3), and matrix metalloproteinase-13 (MMP-13).
Thigh circumference | Baseline and Week 12
  Wrap a flexible measuring tape around the thickest part of the thigh, typically mid-way between the hip and knee. Record the measurement in centimeters or inches.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan